CLINICAL TRIAL: NCT04781348
Title: Efficacy of Platelet Rich Plasma Injection Plus Fat Grafting as Compared to Fat Grafting Alone on Burn Scar by Using Vancouver Scar Scale
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Nasreen Bano, Dr., Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1957
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Burn
Keywords: Platelet-rich plasma; Fat grafting; Efficacy; wound healing; Burns scar; Regeneration
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Group-I: will receive only fat grafting; Group-II: will receive Platelet Rich Plasma and fat grafting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma and fat grafting (Experimental): Group will receive Platelet Rich Plasma plus fat grafting
  Interventions: Procedure: Platelet Rich Plasma plus fat grafting
- Fat grafting (Experimental): Group will receive only fat grafting
  Interventions: Procedure: Platelet Rich Plasma plus fat grafting

INTERVENTIONS:
Procedure: Platelet Rich Plasma plus fat grafting — The study participants fulfilling the inclusion criteria giving consent will be randomly divided into two groups, one group will receive only fat grafting whereas another group will receive Platelet Rich Plasma plus fat grafting.

SUMMARY:
Background: - Burn injuries always leave behind some permanent marks on the body of a victim. For the treatment of these scars, digital photography along with scar scales instrument are an important instrument for the patient's evaluation and finally for the follow-up of scars. Clinical evaluation of the patient after the use of Platelet concentration that it is a beneficial treatment which affects both on hard and soft tissues healing because of having growth factors deposited in PRP. Therefore, it can be used as an alternative to surgery which promotes safe and natural healing in such patients.

Objectives: -

1. To determine the efficacy of Platelet Rich Plasma plus fat grafting as compared to fat grafting alone on the Vancouver scar scale.

Methodology: - An experimental controlled comparison trial study will be done on burn patients, admitted for recovery at the Plastic surgery department, Civil Hospital Karachi after the approval of the scientific committee and Institutional review board of Dow University of Health Sciences, Karachi. The study participants fulfilling the inclusion criteria giving consent will be randomly divided into two groups, one group will receive only fat grafting whereas another group will receive Platelet Rich Plasma plus fat grafting. The sample size of the study will be 52(26 in each group). Both the groups will be followed initially for 15 days of two visits then monthly two visits and finally after 6 months. Assessment of scar with Vancouver Scars Scale (VSS) will be done. The association of the PRP plus fat cells group and control group will be done by applying Chi-square statistical test. P-Value will be set for statistical significance level at <0.05.

DETAILED DESCRIPTION:
OBJECTIVE:

1. To determine the Efficacy of platelet rich plasma injection (PRP) plus fat grafting as compared to fat grafting alone on burn scar by using Vancouver Scar Scale.

HYPOTHESIS:

Null hypothesis:

There is no difference between the effect of Platelet-rich plasma (PRP) plus fat grafting and only fat grafting on the burn scar.

Alternate hypothesis:

There is a difference between the effect and adverse recovery findings of Platelet-rich plasma (PRP) plus fat grafting and only fat grafting on burn scar.

OPERATIONAL DEFINITIONS:

Platelet Rich Plasma (PRP): - Platelet-rich plasma is a blood product that has been enriched with platelets, as a concentrated source of autologous platelets. PRP contains several growth factors and other cytokines that stimulate the healing of bone and soft tissue.

Fat Grafting: - It's a purification process in which fat can be removed from different parts of the body and injected on the face and other areas of the body through a gentle harvesting technique.

Burn Scars: - Burn scars are the scars developed on any part of the body due to burning whatever cause which is depressed, raised, shiny, smooth, or rough, or darker than natural skin and maybe thicker and tougher than normal skin.

METHODOLOGY:

Setting:

Plastic Surgery Department, Civil Hospital Karachi

Study design:

This will be a randomized control trial (RCT) study.

Interventions:

Group-I: will receive only fat grafting Group-II: will receive Platelet Rich Plasma plus fat grafting

Duration:

6 months after the approval of synopsis by the authorizes

Sample size:

The sample size was calculated by Open Epi online sample size software version 3.0. Take fat grafting and PRP, 70% maintenance of contour restoring as compared to only 31% of controls with fat grafting alone 7, 80% of power and 95 confidence levels. The total calculated sample size was 52. After randomization in 8 block with size of 8. we will take 64 (34 in each group).

Block Randomization:

Principal investigator will provide treatments to the both groups. Sixty-six subjects (33 in each group) will be randomizing in 8 block with size of 8 in two treatments group by using online web page sealedenvelope/ create a randomization list. The group I will be treated with fat grafting only from recipient to donor site. Group II will be treated with Platelet-rich plasma plus fat grafting. Both the groups will be followed initially for 15 days of two visits then monthly two visits and finally after 6 months to see if there are any differences between them in outcome (burn scare).

Reference: Create a blocked randomization list | Sealed Envelope, 2021

Inclusion criteria:

1. All the buns patients of either age or sex coming with burn scar for plastic surgery.
2. Give consent for this study
3. Aesthetically not pleasant
4. Exposed body parts
5. Mature scar Exclusion criteria

1. Immature scar 2. Systematic illness. 3. Sepsis 4. Psychiatric illness. 5. Pregnant women

Data collection procedure:

Before starting the project, the approval of the scientific Postgraduate committee and permission from the Institutional Review Board will be taken. All the patients who fulfill the inclusion criteria will be selected for this study. Written consent of the patient will also be taken. Then the patients will be divided into two parts on a random selection basis. The group I will be treated with fat grafting only from recipient to donor site. Group II will be treated with Platelet-rich plasma plus fat grafting. The fat cells will be prepared by Coleman's technique 11. The Platelet Rich Plasma (PRP) will be prepared from (9 - 18 ml). Whole blood of the same person with centrifugation of 3000 (RPm x 3min) with anti-coagulant Citrate Phosphorus Dextrose Adenine-I (CPDA-I) and 4000 (RPm x 15 min) with Calcium Chloride for activation of platelets and normal saline to resolve-centrifugation effect.

This will be done by the highly qualifies pathologist of Dow University of Health Sciences free of cost. Both the groups will be followed initially for 15 days of two visits then monthly two visits and finally after 6 months. Assessment of scar with Vancouver Scars Scale (VSS) will be done. 16

Data analysis procedure:

The collected data will be analyzed through the Statistical Package for the Social Sciences version 20.0. The qualitative variables gender, size, and shape of scare and clinical changes will be presented in frequencies and percentages whereas quantitative variables like age, size of a scare, duration, and assessment of scar with (VSS) Vancouver scare scale will be evaluated through mean ± Standard deviation. The scar will be asses with the Vancouver Scars Scale (VSS) 16. Chi-square statistical test will be applied to assess the difference between the group. P-Value will be set for statistical significance level at <0.05. Efficacy of Platelet Rich Plasma Injection along with fat grafting as compared to fat grafting alone on burn scar in patients of plastic surgery ward of a tertiary care hospital of Karachi.

ELIGIBILITY:
Inclusion Criteria:

1. All the buns patients of either age or sex coming with burn scar for plastic surgery.
2. Give consent for this study
3. Aesthetically not pleasant
4. Exposed body parts
5. Mature scar

Exclusion Criteria:

1. Immature scar
2. Systematic illness.
3. Sepsis
4. Psychiatric illness.
5. Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change in scar | Both the groups will be followed initially for 15 days of two visits then monthly two visits and finally after 6 months.
  Assessment of scar with Vancouver Scars Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic Surgery Department, Civil Hospital Karachi (CHK), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendinelli P, Matteucci E, Dogliotti G, Corsi MM, Banfi G, Maroni P, Desiderio MA. Molecular basis of anti-inflammatory action of platelet-rich plasma on human chondrocytes: mechanisms of NF-kappaB inhibition via HGF. J Cell Physiol. 2010 Nov;225(3):757-66. doi: 10.1002/jcp.22274. PMID 20568106
- [Background] Nakamura S, Ishihara M, Takikawa M, Murakami K, Kishimoto S, Nakamura S, Yanagibayashi S, Kubo S, Yamamoto N, Kiyosawa T. Platelet-rich plasma (PRP) promotes survival of fat-grafts in rats. Ann Plast Surg. 2010 Jul;65(1):101-6. doi: 10.1097/SAP.0b013e3181b0273c. PMID 20548232
- [Background] Cervelli V, Gentile P, Scioli MG, Grimaldi M, Casciani CU, Spagnoli LG, Orlandi A. Application of platelet-rich plasma in plastic surgery: clinical and in vitro evaluation. Tissue Eng Part C Methods. 2009 Dec;15(4):625-34. doi: 10.1089/ten.TEC.2008.0518. PMID 19231923
- [Background] Cervelli V, Gentile P, De Angelis B, Calabrese C, Di Stefani A, Scioli MG, Curcio BC, Felici M, Orlandi A. Application of enhanced stromal vascular fraction and fat grafting mixed with PRP in post-traumatic lower extremity ulcers. Stem Cell Res. 2011 Mar;6(2):103-11. doi: 10.1016/j.scr.2010.11.003. Epub 2010 Nov 30. PMID 21195687
- [Background] Man D, Plosker H, Winland-Brown JE. The use of autologous platelet-rich plasma (platelet gel) and autologous platelet-poor plasma (fibrin glue) in cosmetic surgery. Plast Reconstr Surg. 2001 Jan;107(1):229-37; discussion 238-9. doi: 10.1097/00006534-200101000-00037. PMID 11176628
- [Background] Chandarana S, Fung K, Franklin JH, Kotylak T, Matic DB, Yoo J. Effect of autologous platelet adhesives on dermal fat graft resorption following reconstruction of a superficial parotidectomy defect: a double-blinded prospective trial. Head Neck. 2009 Apr;31(4):521-30. doi: 10.1002/hed.20999. PMID 19156832
- [Result] Brusselaers N, Pirayesh A, Hoeksema H, Verbelen J, Blot S, Monstrey S. Burn scar assessment: a systematic review of different scar scales. J Surg Res. 2010 Nov;164(1):e115-23. doi: 10.1016/j.jss.2010.05.056. Epub 2010 Jun 16. PMID 20828761
- [Result] Jin R, Zhang L, Zhang YG. Does platelet-rich plasma enhance the survival of grafted fat? An update review. Int J Clin Exp Med. 2013 Apr 12;6(4):252-8. Print 2013. PMID 23641301